CLINICAL TRIAL: NCT06801275
Title: The Effect of Number of Showers With 4% Chlorhexidine Gluconate Before Lumbar Disc Herniation Surgery on Prevention of Postoperative Surgical Site Infections: A Single-Blind Randomized Controlled Trial
Brief Title: The Effect of Number of Showers With 4% Chlorhexidine Gluconate on Prevention of Surgical Site Infections
Acronym: SSI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Araz ASKEROĞLU, Assoc. Prof. D., Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20240703591; 2024-116 (Other Grant/Funding Number: Çanakkale Onsekiz Mart University)
Record Dates: First submitted 2025-01-08; First posted 2025-01-30 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Surgical Site Infections; Lumbar Disc Herniation
Keywords: surgical site infections; 4% Chlorhexidine Gluconate
MeSH Terms: conditions — Surgical Wound Infection; Intervertebral Disc Displacement | interventions — chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: Patients to be included in the study will be assigned to experiment-1 or experiment-2 groups by simple randomisation. Routine treatment and care processes in the clinic will be continued for both groups of patients. Experiment 1 group patients will be showered with 4% chlorhexidine gluconate once on the preoperative night. In the experimental group 2 patients, they will be provided to take a shower with 4% chlorhexidine gluconate twice, once on the preoperative night and once on the morning of the operation, by rubbing the waist area for 10 minutes. the effect of the intervention will be evaluated in the postoperative period.
Who Masked: Participant
Masking Description: participants will not know which experimental group they are in
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The effect of 1 shower with 4% chlorhexidine gluconate on surgical site infections (Experimental): Patients will be showered with 4% chlorhexidine gluconate 1 time on the night before surgery.
  Interventions: Other: 1 shower with 4% chlorhexidine gluconate
- The effect of 2 shower with 4% chlorhexidine gluconate on surgical site infections (Other): patients will be provided to shower with 4% chlorhexidine gluconate twice, the night before and the morning of the operation.
  Interventions: Other: 2 shower with 4% chlorhexidine gluconate

INTERVENTIONS:
Other: 1 shower with 4% chlorhexidine gluconate — Comparison of the effect of showering once with 4% Chlorhexidine Gluconate before lumbar disc herniation surgery on surgical site infections
  Other Names: They will be provided to shower with 4% chlorhexidine gluconate once on the night before surgery.
  Arms: The effect of 1 shower with 4% chlorhexidine gluconate on surgical site infections
Other: 2 shower with 4% chlorhexidine gluconate — Comparison of the effect of showering twice with 4% Chlorhexidine Gluconate before lumbar disc herniation surgery on surgical site infections
  Other Names: showering with 4% chlorhexidine gluconate twice, the night before and the morning of surgery
  Arms: The effect of 2 shower with 4% chlorhexidine gluconate on surgical site infections

SUMMARY:
Surgical site infections (SSIs) are the most common type of nosocomial infection in surgical departments.

Although lumbar disc herniation (LDH), which is one of the common cases in neurosurgery, is a serious problem affecting postoperative SSI, morbidity and mortality, there are not enough studies on its prevention in the literature.

In the literature, there are studies on showering with chlorhexidine or other antiseptic solutions in the preoperative period to prevent SSI, but there is no study on whether the number of showers performed in the preoperative period is effective on SSI.

In this study, the effect of showering with 4% chlorhexidine gluconate before lumbar disc herniation surgery on postoperative surgical site infections will be examined. It is aimed to compare the effect of douching with 4% Chlorhexidine Gluconate before lumbar disc hernia surgery on surgical site infections. Since there are not enough studies in the literature, this study is an innovative study. In this study, it is thought that washing the surgical site with antiseptic soap containing 4% Chlorhexidine Gluconate before LDH surgery will have an effect on surgical site infections.

DETAILED DESCRIPTION:
Lumbar disc herniation surgery is performed in two ways: open discectomy and microdiscectomy. In open discectomy, the skin incision is made large enough to expose the lamina and to create an area where the retractor can work with the naked eye. After the lamina is exposed, the correct distance is determined by feeling the sacrum with the fingers. Scopy assistance may be required in suspicious cases. Bone tissue is removed from the lamina to the beginning of the ligamentum flavum without damaging the facet joints. Then the ligament is removed and discectomy is performed by pushing the dura and nerve root inwards. In microdiscectomy, a smaller incision (1.5-2 cm) is made. Special retractors or tubes are inserted. Partial hemilaminotomy and discectomy are performed using microscope and microsurgical instruments.

Although the incidence of SSI after LDH surgery is not known with certainty, patients usually have various potential risk factors for CAI such as advanced age, malnutrition due to loss of appetite, and steroid use. All surgical patients are at risk for developing SSI. For patients, SSI can cause pain and discomfort, financial losses, and impaired quality of life. These infections can lead from a simple incision site abscess with purulent discharge to a complex infection that can contribute to a life-threatening condition and possible morbidity. Therefore, accurate monitoring of SSI and confirmation of the diagnosis of SSI are very important and vital for patients.

The main causative microorganisms of SSI in the preoperative period are gram-positive cocci, which are common bacterial colonies of the skin. Therefore, although WHO recommends showering with normal or antiseptic soap before surgical intervention, it is thought that the use of antiseptic soap will be more effective to destroy a larger number of skin pathogens both before and during surgical intervention.. For this reason, it was deemed appropriate to wash the surgical areas of the patients with antiseptic soap containing 4% chlorhexidine gluconate before surgery.

In the literature, there are studies showing that many factors related to the perioperative process and surgical procedure increase the risk of developing SSI. Among these, there are studies showing that bathing with an antimicrobial agent before surgical intervention reduces the overall bacterial load in the skin's own flora, thus reducing the risk of SSI.

Although there are evidence-based recommendations and some improved care practices to prevent SSI in the literatüre, there is no standardised practice with proven efficacy today. This study is a randomised controlled experimental design and requires a team approach consisting of physicians and nurses in line with the existing evidence recommendations. Therefore, it is thought that showering the operation area with antiseptic soap containing 4% Chlorhexidine Gluconate before lumbar disc herniation surgery will be effective in reducing SSI.

ELIGIBILITY:
Inclusion Criteria:

* to communicate verbally

Exclusion Criteria:

* Patients with diabetes mellitus side disease, pylolidal cyst surgery, any surgical history from the lumbar region and patients who will undergo lumbar disc hernia stabilisation surgery will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
surgical site infection | 30 days following surgical intervention
  Following the surgical intervention, the surgical site will be monitored for purulent discharge, abscess or cellulitis for 30 days. The patients will be followed up by the investigator and the specialist physician in the clinic until discharge and by the investigator after discharge. In the postoperative period, purulent discharge, abscess or cellulitis that develops in the surgical site within 30 days following the surgical intervention will be defined as SSI with the approval of the specialist physician.

CONTACTS AND LOCATIONS:
Overall Officials: araz askeroğlu, Study Director — çanakkale on sekiz mart university
Locations (2):
- Turkey (Türkiye) (2):
  - Çanakkale on Sekiz Mart University, Çanakkale, Merkez
  - Çanakkale on Sekiz Mart Üniversity, Çanakkale, Merkez

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sway A, Solomkin JS, Pittet D, Kilpatrick C. Methodology and Background for the World Health Organization Global Guidelines on the Prevention of Surgical Site Infection. Surg Infect (Larchmt). 2018 Jan;19(1):33-39. doi: 10.1089/sur.2017.076. Epub 2017 May 4. PMID 28472604
- [Background] Young H, Bliss R, Carey JC, Price CS. Beyond core measures: identifying modifiable risk factors for prevention of surgical site infection after elective total abdominal hysterectomy. Surg Infect (Larchmt). 2011 Dec;12(6):491-6. doi: 10.1089/sur.2010.103. Epub 2011 Dec 5. PMID 22142313
- [Background] McClelland S 3rd, Hall WA. Postoperative central nervous system infection: incidence and associated factors in 2111 neurosurgical procedures. Clin Infect Dis. 2007 Jul 1;45(1):55-9. doi: 10.1086/518580. Epub 2007 May 21. PMID 17554701
- [Background] Abode-Iyamah KO, Chiang HY, Winslow N, Park B, Zanaty M, Dlouhy BJ, Flouty OE, Rasmussen ZD, Herwaldt LA, Greenlee JD. Risk factors for surgical site infections and assessment of vancomycin powder as a preventive measure in patients undergoing first-time cranioplasty. J Neurosurg. 2018 Apr;128(4):1241-1249. doi: 10.3171/2016.12.JNS161967. Epub 2017 May 12. PMID 28498056
- [Background] Aldrich A, Kuss MA, Duan B, Kielian T. 3D Bioprinted Scaffolds Containing Viable Macrophages and Antibiotics Promote Clearance of Staphylococcus aureus Craniotomy-Associated Biofilm Infection. ACS Appl Mater Interfaces. 2019 Apr 3;11(13):12298-12307. doi: 10.1021/acsami.9b00264. Epub 2019 Mar 21. PMID 30855125
- [Background] AORN. (2014). Preoperative Standards and Recommended Practices. Denver, CO: AORN, pp. 445-463.
- [Background] Berrios-Torres SI, Umscheid CA, Bratzler DW, Leas B, Stone EC, Kelz RR, Reinke CE, Morgan S, Solomkin JS, Mazuski JE, Dellinger EP, Itani KMF, Berbari EF, Segreti J, Parvizi J, Blanchard J, Allen G, Kluytmans JAJW, Donlan R, Schecter WP; Healthcare Infection Control Practices Advisory Committee. Centers for Disease Control and Prevention Guideline for the Prevention of Surgical Site Infection, 2017. JAMA Surg. 2017 Aug 1;152(8):784-791. doi: 10.1001/jamasurg.2017.0904. PMID 28467526
- [Background] Damkliang J, Considine J, Kent B, Street M. Nurses' perceptions of using an evidence-based care bundle for initial emergency nursing management of patients with severe traumatic brain injury: A qualitative study. Int Emerg Nurs. 2015 Oct;23(4):299-305. doi: 10.1016/j.ienj.2015.04.004. Epub 2015 Jun 3. PMID 26049810
- [Background] Edmiston CE Jr, Leaper D. Should preoperative showering or cleansing with chlorhexidine gluconate (CHG) be part of the surgical care bundle to prevent surgical site infection? J Infect Prev. 2017 Nov;18(6):311-314. doi: 10.1177/1757177417714873. Epub 2017 Jul 26. PMID 29344102
- [Background] Liu H, Dong X, Yin Y, Chen Z, Zhang J. Reduction of Surgical Site Infections After Cranioplasty With Perioperative Bundle. J Craniofac Surg. 2017 Sep;28(6):1408-1412. doi: 10.1097/SCS.0000000000003650. PMID 28692506